CLINICAL TRIAL: NCT02079155
Title: Prospective Single-Center Randomized Study of Robotic Athermal Nerve-Sparing Radical Prostatectomy: Laparoendoscopic Single-Site Versus Standard Approach
Brief Title: Robotic Athermal Nerve-Sparing Radical Prostatectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research Cancelled
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE12811; NCI-2014-00393 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE12811 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Stage I Prostate Cancer; Stage IIA Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (RALP) (Active Comparator): Patients undergo standard RALP.
  Interventions: Procedure: robot-assisted laparoscopic surgery; Other: laboratory biomarker analysis; Other: quality-of-life assessment; Other: questionnaire administration
- Arm II (R-LESS RP) (Experimental): Patients undergo R-LESS RP.
  Interventions: Procedure: robot-assisted laparoscopic surgery; Other: laboratory biomarker analysis; Other: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Procedure: robot-assisted laparoscopic surgery — Undergo RALP
  Arms: Arm I (RALP)
Procedure: robot-assisted laparoscopic surgery — Undergo R-LESS RP
  Arms: Arm II (R-LESS RP)
Other: laboratory biomarker analysis — Correlative studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized clinical trial compares a recently developed technique, called robotic laparoendoscopic single-site radical prostatectomy (R-LESS RP), to the current standard of robotic technique for prostate cancer, robot-assisted laparoscopic prostatectomy (RALP) in treating patients with newly diagnosed, locally confined prostate cancer. Both procedures are types of robotic radical prostatectomy, or the robot-assisted removal of the prostate though a small incision in the belly. In the standard approach, 4-5 small (1-2 cm) incisions are made in the lower abdomen to allow the insertion of robotic instruments. In the R-LESS technique, all instruments are inserted through a single incision. R-LESS RP is less invasive than RALP and may leave a smaller scar and cause less pain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate pain and analgesic requirement of R-LESS RP compared to standard RALP.

SECONDARY OBJECTIVES:

I. Time to oral intake. II. Time to resume ambulation. III. Hospital stay, counted in whole days from the day of surgery to the day of discharge.

IV. Perioperative parameters, including: operative time (defined as time elapsed from skin incision to placement of the final skin suture); estimated blood loss; additional ports; conversion to standard RALP (in R-LESS RP patients), or laparoscopic, or open surgery; length of stay.

V. Intraoperative complications. VI. Postoperative complications, recorded according to the Clavien classification.

VII. Body image perception, measured using the body image questionnaire (BIQ). VIII. Scar evaluation (at suture removal and at 6 month) by using a validated assessment tool, the Patient and Observer Scar Assessment Scale.

IX. Health related quality of life, measured as patients' perception of functioning, disability, and well-being related to the following eight concepts: physical functioning, role limitations caused by physical health problems, bodily pain, general health, vitality, social functioning, role limitation caused by emotional problems, and mental health.

X. Urinary continence, assessing the number of pads used daily. XI. Erectile Function, assessed by the International Index of Erectile Function (IIEF-5).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo standard RALP.

ARM II: Patients undergo R-LESS RP.

After completion of study treatment, patients are followed up periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a biopsy proven newly diagnosed locally confined, stage T1a, T2a or T2b prostate cancer
* Judged by the study doctor to be a suitable candidate for a radical prostatectomy
* Serum prostate specific antigen equal to or less than 10 ng/mL
* Gleason score equal to or less than 7
* Life expectancy greater than 10 years
* Prostate size on trans-rectal ultrasound (TRUS) measurement less than 50 grams
* Favorable operative risk defined as American Society of Anesthesiology Score (ASA score) =< 3
* Ability to understand and the willingness to sign a written informed consent document or have a surrogate with the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients with any prior pelvic surgery
* Patients with prior history of pelvic fractures or hip replacement
* Large pelvic or intra-abdominal masses
* Any condition or history of illness or surgery that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient (e.g. significant cardiovascular conditions)
* Poor surgical risk (defined as American Society of Anesthesiology Score > 3)
* Active infection
* Uncorrected coagulopathy
* Body mass index equal to or greater than 35

Ages: 35 Years to 72 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mean pain score, evaluated with the visual analog pain score (VAPS) | Up to 1 year
  Compared using the Mann-Whitney U test as appropriate.
Mean analgesic consumption, obtained from medical charts and reported as units of parenteral morphine equivalents (mg) | Up to 1 month
  Compared using the Mann-Whitney U test as appropriate.

SECONDARY OUTCOMES:
Time to oral intake | Up to 1 year
  Compared using the Mann-Whitney U test as appropriate.
Time to resume ambulation | Up to 1 year
  Compared using the Mann-Whitney U test as appropriate.
Length of hospital stay, counted in whole days from the day of surgery to the day of discharge | Up to 3 days
  Compared using the Mann-Whitney U test as appropriate.
Operative time, defined as time elapsed from skin incision to placement of the final skin suture | Day 1
  Compared using the Mann-Whitney U test as appropriate.
Estimated blood loss during surgery | Day 1
  Compared using the Mann-Whitney U test as appropriate.
Additional ports during surgery | Day 1
  Compared using the Mann-Whitney U test as appropriate.
Incidence of conversion to standard RALP, laparoscopic, or open surgery in R-LESS RP patients | Day 1
  Compared by means of Fisher's exact test.
Incidence of intraoperative complications | Day 1
  Compared using the Mann-Whitney U test as appropriate.
Incidence of postoperative complications, recorded according to the Clavien classification | Up to 1 year
  Compared using the Mann-Whitney U test as appropriate.
Body image perception, measured using the BIQ | Up to 1 year
  Compared using the Mann-Whitney U test as appropriate. The BIQ consists of two scales: the body image scale, which assesses attitudes to bodily appearance and consists of five questions (score 5-20), and the cosmetic scale which assesses degree of satisfaction with the appearance of the scare and consists of three questions (score 3-24).
Scar evaluation, assessed using the Patient and Observer Scar Assessment Scale | Up to 1 year
  Compared using the Mann-Whitney U test as appropriate. Assessed at suture removal and at 6 months. The Patient and Observer Scar Assessment Scale consists of two scales: the observer scale and the patient scale. Both scales contain 6 items that are scored numerically. Each of the six items on both scales has a 10-step score, with 10 indicating the worst imaginable scar or sensation. The total score of both scales consists of adding the scores of each of the six items (range, 6 to 60). The lowest score, 6, reflects normal skin, whereas the highest score, 60, reflects the worst imaginable scar.
Health related quality of life, measured as patients' perception of functioning, disability, and well-being | Up to 1 year
  Compared using the Mann-Whitney U test as appropriate. Patients' perception of functioning, disability, and well-being will be measured related to the following eight concepts: physical functioning, role limitations cause by physical health problems, bodily pain, general health, vitality, social functioning, role limitation caused by emotional problems, and mental health.
Urinary continence, assessed by the number of pads used daily | Up to 12 months
  Compared using the Mann-Whitney U test as appropriate. Evaluated at 1, 3, 6, and 12 months after the procedure.
Erectile function, assessed by the IIEF-5 | Up to 12 months
  Compared using the Mann-Whitney U test as appropriate. Evaluated once in preoperative period and at 1, 3, 6, and 12 months after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Kaouk, Principal Investigator — Case Comprehensive Cancer Center